CLINICAL TRIAL: NCT06681298
Title: A Multi-center, Two-arm, Phase 2 Clinical Study on the Perioperative Treatment of HER2-positive Resectable Esophagogastric Junctional Adenocarcinoma With Nabulimab Combined With FLOT and Trastuzumab VS FLOT Combined With Trastuzumab
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: xiaohua li (Other)
Responsible Party: Sponsor-Investigator, xiaohua li, professor, Xijing Hospital of Digestive Diseases
Organization: Xijing Hospital of Digestive Diseases (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20242180-C-1
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Adenocarcinoma of the Esophagogastric Junction; Perioperative Period
Keywords: Nivolumab; adenocarcinoma of the esophagogastric junction; FLOT
MeSH Terms: interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nivolumab group (Experimental): Preoperative nabuliumab combined with FLOT and trastuzumab + surgical treatment + postoperative nabuliumab combined with FLOT and trastuzumab. There were 4 cycles before and after surgery, one cycle every 2 weeks. The specific administration was: docetaxel 50mg/m2 iv,d1, oxaliplatin 85mg/m2 iv,d1, calcium leucovorin 200mg/m2 iv,d1,5-FU 2600mg/m2 iv,d1, infusion 24h; Nebulizumab 240mg iv,d2, 30 minutes per intravenous infusion, trastuzumab 4mg/kg iv,d2 (load dose 6mg /kg).
  Interventions: Drug: The experimental group received Nivolumab
- Control group (Active Comparator): The control group was treated with preoperative FLOT combined with trastuzumab + surgical treatment + postoperative FLOT combined with trastuzumab. Preoperative and postoperative cycles were 4 in both groups, with one cycle every 2 weeks. Specific administration was as follows: Docetaxel 50mg/m2 iv,d1, oxaliplatin 85mg/m2 iv,d1, calcium leucovorin 200mg/m2 iv,d1,5-FU 2600mg/m2 iv,d1, infusion 24h; Trastuzumab 4mg/kg iv,d2 (load dose 6mg /kg).
  Interventions: Drug: The experimental group received Nivolumab

INTERVENTIONS:
Drug: The experimental group received Nivolumab — Trastuzumab and the FLOT chemotherapy regimen are clearly recommended by guidelines, whereas Nivolumab is currently requiring further research validation.
  Other Names: Trastuzumab; FLOT

SUMMARY:
Patients with Her2+ resectable gastroesophageal conjunctive adenocarcinoma were randomly divided into observation group and control group. The observation group received preoperative nabuliumab combined with FLOT and trastuzumab + surgical treatment + postoperative nabuliumab combined with FLOT and trastuzumab. The control group was treated with preoperative FLOT combined with trastuzumab + surgical treatment + postoperative FLOT combined with trastuzumab. 4 cycles were performed before and after surgery in both groups, with one cycle every 2 weeks. The specific administration was docetaxel 50mg/m2 iv,d1, oxaliplatin 85mg/m2 iv,d1, calcium leucovorin 200mg/m2 iv,d1,5-FU 2600mg/m2 iv,d1, infusion 24h; Nebulizumab 240mg iv,d2, 30 minutes per intravenous infusion, trastuzumab 4mg/kg iv,d2 (load dose 6mg /kg). Surgical treatment was evaluated by the investigator within 3-4 weeks after the last dosing. After 4 cycles of adjuvant therapy, the observation group received nebuliumab combined with trastuzumab, while the control group received maintenance therapy with trastuzumab. Both groups received 10 cycles, one cycle every 2 weeks. The specific administration was as follows: nebuliuzumab 240mg iv,d1, 30 minutes per intravenous infusion; Trastuzumab 4mg/kg intravenously.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized controlled clinical study. A total of 36 patients with locally advanced esophagogastric conjoint adenocarcinoma without any treatment and resection were included in this study. After signing informed consent and meeting the screening criteria, a total of 36 patients were randomized into the observation group and the control group (18 cases and 18 cases, respectively) without blindness. Other participants include the Second Affiliated Hospital of Air Force Medical University, Henan Provincial People's Hospital, Cancer Hospital of Tianjin Medical University, Zhongshan Hospital Affiliated to Shanghai Fudan University, and the First Affiliated Hospital of Xi 'an Jiaotong University. The research groups were as follows: patients with resectable gastroesophageal conjunctive adenocarcinoma were randomly divided into observation group and control group. The observation group received preoperative nabuliumab combined with FLOT and trastuzumab + surgical treatment + postoperative nabuliumab combined with FLOT and trastuzumab. The control group was treated with preoperative FLOT combined with trastuzumab + surgical treatment + postoperative FLOT combined with trastuall Zumab. Preoperative and postoperative cycles were 4 in both groups, with one cycle every 2 weeks. Specific administration was as follows: Docetaxel 50mg/m2 iv,d1, oxaliplatin 85mg/m2 iv,d1, calcium leucovorin 200mg/m2 iv,d1,5-FU 2600mg/m2 iv,d1, infusion 24h; Nebulizumab 240mg iv,d2, 30 minutes per intravenous infusion, trastuzumab 4mg/kg iv,d2 (load dose 6mg /kg). At 3-4 weeks after the completion of the last dosing cycle, the efficacy of neoadjuvant therapy and the possibility of radical resection were evaluated in combination with preoperative imaging examination, and radical surgical treatment was performed. After the operation, the investigator will determine whether to carry out adjuvant treatment and choose the appropriate treatment plan (the first treatment should start from 3-6W after the operation and should not exceed 3 months). After 4 cycles of adjuvant therapy, the observation group was treated with nebuliumab combined with trastuzumab, and the control group was treated with trastuzumab maintenance therapy, with 10 cycles for each The specific administration was as follows: 240mg iv,d1, intravenous infusion for 30 minutes each time; Trastuzumab 4mg/kg intravenously. Resection of esophagogastric junction carcinoma was performed based on the 2023 Chinese Society of Clinical Oncology (CSCO) Guidelines for the Diagnosis and treatment of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old;
2. esophagogastric junction adenocarcinoma (including Siewert type I, Siewert type II, and Siewert type III) with histopathologic or cytological confirmation of HER2-positive (defined as positive immunohistochemical [IHC] greater than or equal to 2+ and fluorescence in situ hybridization [FISH]);
3. The cTNM stages were cT3-4a, N+, M0 according to endoscopic ultrasound or enhanced CT/MRI scanning (combined with ultrasonic gastroscopy and diagnostic laparoscopic exploration if necessary) (refer to the 8th edition AJCCTNM staging system), and the lesions were resected as assessed by the investigator;
4. Expected survival time > 6 months;
5. ECOG PS score 0 or 1;
6. PD-L1 does not require;
7. No prior treatment;
8. Hematological indexes were basically normal: white blood cell count ≥4×109/L; Absolute neutrophil count ≥1.5×109/L; Platelet ≥100×109/L; Hemoglobin ≥ 90 g/Lg/L;
9. Basically normal renal function: serum creatinine ≤1.5×ULN or creatinine clearance (CrCl)>60 mL/min(using the Cockcroft-Gault formula);
10. Basically normal liver function: serum total bilirubin ≤1.5×ULN; Aspartate aminotransferase (AST) ≤2.5×ULN; Alanine aminotransferase (ALT) ≤2.5×ULN;
11. Female patients must have a negative urine pregnancy test before the start of the study (not applicable to patients with bilateral oophorectomy and/or hysterectomy or postmenopausal patients)
12. Sign written informed consent.

Exclusion Criteria:

* (1) No efficacy and/or safety evaluation has been performed; (2) The investigator believes that the patient is not suitable to continue (reasons for withdrawal should be recorded) (3) The patient requested that the trial be terminated; (4) Serious violation of protocol: participating in this study while using other anti-tumor drugs and/or modern Chinese medicine preparations with anti-cancer indications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | 30 days
  Pathological complete response rate refers to the proportion of primary tumor sites and surgical specimens with no viable tumor cells (ypT0N0) in all resected lymph nodes to the total number of patients evaluated centrally by the study pathologist

SECONDARY OUTCOMES:
Objective response rate (ORR) | 30 days
  Objective response rate (ORR) : ORR is the proportion of subjects who achieved partial and complete response on imaging assessment (RECIST v1.1) after the end of neoadjuvant therapy
Progression-free survival (PFS) | 1,3,5 years
  Progression-free survival (PFS) : PFS is the time from the date of enrollment in the study to the date of death from all causes
Overall survival (OS) | 1,3,5 years
  Overall survival (OS) : OS is the amount of time a patient can survive treatment without dying from any condition
Major pathological response rate (MPR) | 30 days
  Major pathological response rate (MPR) : MPR refers to the proportion of patients with residual tumor cells < 10% after surgery to determine the pathological status of the primary lesion
Duration of response (DOR) | 5 years
  Duration of response (DOR) : The DOR is the time from the first response until disease progression is first recorded or death occurs
Adverse Event Rate (AE) | 5 years
  Adverse Event Rate (AE) : Any adverse events that may be related to the investigational drug that occur while receiving neoadjuvant therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ruiqi Gao, Principal Investigator — Department of Gastrointestinal Surgery, Xijing Hospital, Fourth Military Medical University
Locations (1):
- The First Affiliated Hospital of the Air Force Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Share in the form of an article or email
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: start date :2024-5-1; finish date:2029-5-1.
Access Criteria: Share in the form of an article or email(1073297317@qq.com)
URL: https://clinicaltrials.gov